

## Intensive care decision-making, survival and dying well:

How do the experiences of intensive care patients and their end-of-life wishes affect their willingness to accept intensive care treatment at different chances of survival?

## **Consent Form**

If you are happy to participate, please complete and sign the consent form below

| | Activities | Initials |
|---|---|---|
| 1 | I confirm that I have read the attached information sheet ( <b>Version 4, Date 19/10/2022</b> ) for the above study and have had the opportunity to consider the information and ask questions and had these answered satisfactorily. | |
| 2 | I understand that my participation in the study is voluntary and that I am free to withdraw at any time without giving a reason and without detriment to myself. I understand that it will not be possible to remove my data from the project once it has been anonymised and forms part of the data set. | |
| | I agree to take part on this basis. | |
| | I agree to my GP being informed of my participation in this study. Please provide your GP's address: | |
| 3 | | |
| 4 | I agree to the interviews being audio recorded to enable a transcript of the interview to be produced. The audio recording will be destroyed once the transcription is completed. | |
| 5 | I agree that any data collected, including anonymous quotations from the transcript, may be included in anonymous form in publications/conference presentations and in the final study report. | |
| 6 | I understand that a fully anonymised dataset will be deposited in an open data repository at the end of the project and that any anonymised data collected may be made available to other researchers | |
| 7 | I understand that data collected during the study will be stored securely in line with the University of Manchester data protection policy and that the data may be looked at by individuals from The University of Manchester, regulatory authorities or the NHS Trust, where it is relevant to my taking part in this research to make sure the project is being carried out as planned. This may involve looking at identifiable data but, all individuals involved in auditing and monitoring the study will have a strict duty of confidentiality to me as a research participant. I give permission for these individuals to have access to my data. | |



| 8 | I understand that there may be instances where during the course of the research information is revealed which means the researchers will be obliged to break confidentiality and this has been explained in more detail in the information sheet. |
|---|---|
| 9 | I agree to take part in this study. |

The following activities are optional, you may participate in the research without agreeing to the following:

| 15 | I agree that any personal data collected may be made available to other researchers |
|---|---|
| 16 | I agree that the researchers may contact me in future about other research projects. |
| 17 | I agree that the researchers may retain my contact details in order to provide me with a summary of the findings for this study. |

## **Data Protection**

The personal information we collect and use to conduct this research will be processed in accordance with data protection law as explained in the Participant Information Sheet and the <a href="Privacy Notice for Research Participants">Privacy Notice for Research Participants</a>.

| Name of Participant | Signature | Date |
|-------------------------------------|-----------|------|
| Dr Thomas Donaldson<br>(Researcher) | | |
| Name of the person taking consent | Signature | Date |

Please keep one copy of this form for yourself, and return the original signed copy of this form to the research team in the stamped addressed envelope.